CLINICAL TRIAL: NCT06795906
Title: A Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of AZD8630, Administered Once Daily Via Inhalation, for 2 Weeks, in Adults With Asthma on Medium-to-high Dose Inhaled Corticosteroids and Long-acting Beta-agonists
Brief Title: A Safety, Pharmacokinetic, and Pharmacodynamic Study of Once Daily Inhaled AZD8630 in Adults With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6830C00004
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Asthma
Keywords: Inhaled corticosteroids; Long-acting beta-agonists
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD8630 Dose A (Experimental): Participants will self-administer AZD8630 Dose A daily from Day 1 up to Day 14.
  Interventions: Drug: AZD8630; Device: Saphira device
- Placebo (Placebo Comparator): Participants will self-administer corresponding placebo daily from Day 1 up to Day 14.
  Interventions: Other: Placebo; Device: Saphira device

INTERVENTIONS:
Drug: AZD8630 — AZD8630 will be administered via dry powder inhalation (DPI).
  Arms: AZD8630 Dose A
Other: Placebo — Placebo will be administered via DPI.
  Arms: Placebo
Device: Saphira device — AZD8630 or placebo will be administered to participants via Saphira device.

SUMMARY:
This is a randomised, placebo-controlled, double-blinded, sponsor-unblinded study to assess the safety, pharmacokinetic (PK), and pharmacodynamic (PD) effect of AZD8630 in adult participants with asthma on medium-to-high dose inhaled corticosteroids (ICS) and long-acting beta-agonists (LABA).

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, PK, and PD of AZD8630 compared to placebo in participants with asthma and elevated fractional exhaled nitric oxide (FeNO) on a combination of medium-to-high dose ICS and LABA medications.

The study will comprise of:

* A Screening/Enrollment Period of up to 14 to 28 days before dosing.
* A Treatment Period/End of Treatment Visit. On Day 1, participants will be randomised to AZD8630 or corresponding placebo. Study intervention will be self-administered once daily up to Day 14. Participants will return to the study site for clinical and safety assessments on Day 7 and clinical and safety assessments and PK sampling on Day 14.
* A Follow-up Visit 1 week after last dose.

ELIGIBILITY:
Inclusion Criteria:

1 Participants who have documented physician-diagnosis of asthma for at least 12 months, as evidenced by any of the following:

1. Post-bronchodilator (BD) reversibility of FEV1 ≥ 12% and ≥ 200 milliliters (mL) within 5 years prior to Visit 1, at Visit 1 or
2. Peak expiratory flow (PEF) average daily variability > 10% over a 2-week period within 5 years prior to Visit 1, or
3. Variability of FEV1 > 12% and 200 mL between any 2 clinical visits within 5 years prior to Visit 1, or
4. Positive bronchial challenge test within 5 years prior to Visit 1. A positive test is defined as a fall in FEV1 from pre-challenge of ≥ 20% with standard doses of methacholine or ≥ 5% with standardised hyperventilation, hypertonic saline, or mannitol challenge, or
5. Positive exercise challenge test within 5 years prior to Visit 1. A positive test is defined as a fall in FEV1 of > 10% and > 200 mL from pre-challenge, or
6. Significant increase in lung function after 4 weeks of Inhaled Corticosteroids (ICS) anti-inflammatory treatment within 5 years prior to Visit 1, defined as an increase in FEV1 > 12% and 200 mL (or PEF by > 20%).

   3 Treated with medium or high dose ICS (as per GINA 2023) in combination with long-acting beta-agonists (LABA) (GINA step 4 or 5 therapy); the dose of ICS must be stable for at least 30 days prior to Visit 1. The ICS can be contained within an ICS-LABA fixed-dose combination product.

   - Treatment with additional asthma controller therapies (eg, long-acting muscarinic-agonists) at a stable dose ≥ 30 days prior to Visit 1 is allowed.

   4 Asthma Control Questionnaire-6 (ACQ-6) score in the range 0.75-3 at both screening and randomisation.

   5 Pre-bronchodilator FEV1 ≥ 40%. 6 FeNO ≥ 30 parts per billion (ppb) at both screening and randomisation. 7 At least 70% compliance with usual asthma background medication during the screening period (14 days prior to randomisation) based on the daily asthma ePROs. At least 70% compliance with electronically recorded participant reported outcomes (ePRO) device completion during the screening period (14 days prior to randomisation). This is defined as completing the ePRO any 10 mornings and 10 evenings in the last 14 days prior to randomisation.

   8 Minimum 70% compliance with PEF measurements during the screening period (14 days prior to randomisation). This is defined as performing PEF for any 10 mornings and any 10 evenings in the last 14 days prior to randomisation.

   9 Body mass index (BMI) within the range 18 to 35 kilograms per meter (kg/m2) inclusive and weight at least 45 kg at the time of signing the informed consent.

Exclusion Criteria:

1. Life-threatening asthma defined as a history of significant asthma episode(s) involving intubation, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s).
2. Completed treatment for respiratory infection and/or asthma exacerbation with systemic corticosteroids and/or antibiotics in the 4 weeks prior to Visit 1 or during the screening period.
3. Clinically important pulmonary disease other than asthma; including but not limited to participants with co-existent chronic obstructive pulmonary disease (COPD).
4. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator and could:

   1. Affect the safety of the participant throughout the study.
   2. Influence the findings of the study or the interpretation.
   3. Impede the participant's ability to complete the entire study.
5. Participants who, in the opinion of the investigator, have evidence of active tuberculosis (TB) or are currently on treatment for active or latent TB. Investigation for active or latent TB with interferon gamma release assay (IGRA) and/or chest X-ray should only be considered if deemed clinically indicated by the Principal Investigator.
6. Medical history of or treatment for hepatitis B or hepatitis C, except for cured hepatitis C, as defined by:

   1. Positive test for hepatitis B surface antigen (HBsAg).
   2. Positive test for anti- hepatitis B core antibody (HBc Ab): Participants who test positive for anti-HBc Ab but negative for HBsAg may be enrolled if their hepatitis B virus (HBV) DNA test result is negative.
   3. Positive test for anti-hepatitis C antibody: Participants who test positive for anti-hepatitis C antibody may be enrolled if their hepatitis C viral ribonucleic acid (RNA) test result is negative in the absence of cirrhosis.
7. Participants with known human immunodeficiency virus (HIV) or with a positive HIV test at screening.
8. Any other clinically relevant abnormal findings in laboratory testing including haematology and clinical chemistry, on vital signs, electrocardiogram (ECG), or physical examination between consent and randomisation, that in the opinion of the investigator or medical monitor, might compromise the safety of the participant in the study or interfere with evaluation of the study intervention. Abnormal findings include, but are not limited to:

   1. Alanine aminotransferase/transaminase (ALT) or aspartate aminotransferase/transaminase AST > 2 × upper limit of normal (ULN).
   2. Total bilirubin (TBL) > 1.5 × ULN (unless due to Gilbert's disease).
   3. Evidence of chronic liver disease.
9. Congenital long QT syndrome or prolonged QT corrected for heart rate by Fridericia (QTcF) > 470 ms or history of QT prolongation associated with other medications that required discontinuation of that medication.
10. Current untreated or uncontrolled arrhythmia (eg, multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia). Note: Participants with clinically significant sinus nodal disease/bradycardia or Type 2 second- or third-degree atrioventricular (AV) block can be included if treated with pacemaker.
11. Participants with recent (within 3 months of Visit 1) myocardial infarction, unstable angina pectoris, stroke, percutaneous coronary intervention and coronary artery bypass grafting (within 6 months of Visit 1).
12. Current smokers, former smokers with > 10 pack-years history, or former smokers who stopped smoking < 6 months before Visit 1 (including all forms of tobacco, e-cigarettes (vaping), and other recreational drugs including marijuana).
13. History of current or previous alcohol or drug misuse in the 12 months prior to screening. The use of oral cannabis is permitted.
14. Current diagnosis of cancer or unresectable cancer that has not been in complete remission for at least 5 years prior to Visit 1. Note: Squamous cell and basal cell carcinomas of the skin and cervical carcinoma-in-situ that have been treated and considered cured at the time of enrolment are not exclusionary.
15. History of documented immune complex disease (Type III hypersensitivity reactions) to monoclonal antibody (mAb) administration.
16. History of hypersensitivity or anaphylaxis to any components of AZD8630 formulation.
17. History of anaphylaxis or ongoing clinically important serious allergy, as judged by the investigator, or history of anaphylaxis that required the use of epinephrine/adrenaline or hospitalisation.
18. A helminth parasitic infection diagnosed within 24 weeks of screening that has not been treated or has not responded to standard of care therapy.
19. Use of the following medicines within the specified time before screening:

    1. Treatment with marketed or investigational biologics for asthma or immunological disease within 4 months or a minimum of 5 half-lives, whichever is longer, prior to the screening visit.
    2. Systemic steroids within 4 weeks prior to the screening visit. Note: Intranasal steroid use is permitted, provided that there has been a stable treatment regimen for 4 weeks.
    3. Live, attenuated, or mRNA vaccine in the 4 weeks prior to screening visit.
    4. Any systemic immunosuppressive therapy within 3 months of screening visit until the end of the follow-up period.
    5. Use of allergen immunotherapy within 3 months of screening visit, except for stable maintenance dose allergen-specific immunotherapy started 4 weeks prior to screening visit.
    6. Bronchial thermoplasty in the last 12 months prior to screening visit.
    7. Receipt of immunoglobulin or blood products within 4 weeks prior to screening visit.
20. Participation in another clinical study with a study intervention administered within 5 half-lives or in accordance with local regulations (whichever is longer) prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) and serious adverse events (SAEs) | From Screening (Day -28) to Follow up (Day 21)
  To assess the safety and tolerability of AZD8630 Dose A daily (QD) in participants with asthma on medium-to-high dose ICS and LABA.
Number of adverse events leading to discontinuation (DAEs) | From Day 1 to Day 14
  To assess the safety and tolerability of AZD8630 Dose A QD in participants with asthma on medium-to-high dose ICS and LABA.
Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) | Day 1, Day 14 and Follow up (Day 21)
  To assess the PK of AZD8630 Dose A QD in participants with asthma on medium-to-high dose ICS and LABA.
Maximum observed plasma (peak) drug concentration (Cmax) | Day 1, Day 14 and Follow up (Day 21)
  To assess the PK of AZD8630 Dose A QD in participants with asthma on medium-to-high dose ICS and LABA.

SECONDARY OUTCOMES:
Change from baseline in fractional exhaled nitric oxide (FeNO) at Weeks 1 and 2 | From Screening (Day -28) to Follow up (Day 21)
  To evaluate the PD of AZD8630 Dose A QD in participants with asthma on medium-to-high dose ICS and LABA.
Incidence of anti-drug antibodies (ADAs) in serum | Day 1, Day 14 and Follow up (Day 21)
  To characterise the immunogenicity of AZD8630 Dose A QD in participants with asthma on medium-to-high dose ICS and LABA.
Incidence of AEs and SAEs associated with the Saphira device | Day 1 to Day 14
  To assess the safety and performance of the Saphira device.
Incidence of Saphira device deficiencies (DDs) | Day 1 to Day 14
  To assess the safety and performance of the Saphira device.
Incidence of participant confirmation of dose administration following inhalation | Day 1 to Day 14
  To assess the safety and performance of the Saphira device.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Research Site, Ahrensburg
  - Research Site, Berlin
  - Research Site, Mainz

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/